CLINICAL TRIAL: NCT03190421
Title: The Use of Expanded Quantitative Urinary Culture (EQUC) Versus Standard Culture (SUC) Techniques in the Clinical Care of Women With Symptoms of Urinary Tract Infections.
Brief Title: Expanded Quantitative Urinary Culture (EQUC) vs Standard Culture (SUC) Techniques in the Clinical Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Elizabeth Mueller, M.D., Professor, Loyola University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 209545
Record Dates: First submitted 2017-06-14; First posted 2017-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Intervention Model Description: Expanded Quantitative Urinary Culture (EQUC) versus Standard Culture (SUC) Techniques
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expanded Urinary Culture (EQUC) (Experimental): Participants in this arm will receive the expanded urine culture
  Interventions: Diagnostic Test: Expanded Urinary Culture
- Standard Urine Culture (SUC) (Active Comparator): Participants in this arm will receive the standard urine culture
  Interventions: Diagnostic Test: Standard Urine Culture (SUC)

INTERVENTIONS:
Diagnostic Test: Expanded Urinary Culture — involves the inoculation of 100X (0.1mL) more urine onto diverse types of media (BAP, chocolate agar, colistin and nalidixic acid (CNA) agar, CDC anaerobe 5% BAP) with incubation in more environments and temperatures (5% CO2 at 35°C for 48 h, aerobic conditions at 35°C and 30°C for 48 h, Campy gas mixture (5% O2, 10% CO2, 85% N) or anaerobic conditions at 35°C for 48 h). The level of detection for EQUC is 10 CFU/mL, represented by 1 colony of growth on any of the plates. EQUC is designed to isolate a broad array of Gram-negative and Gram-positive bacteria, including anaerobes and fastidious bacteria that grow slowly.
  Arms: Expanded Urinary Culture (EQUC)
Diagnostic Test: Standard Urine Culture (SUC) — involves inoculation of 0.001 mL of urine onto 5% sheep blood agar plate (BAP) and MacConkey agar plate with the plates being incubated aerobically at 35°C for 24 h. Thus, the level of detection for standard culture is 103 CFU/mL, represented by 1 colony of growth on either plate. Standard culture is designed specifically to grow Gram-negative rods, especially UPEC.
  Arms: Standard Urine Culture (SUC)

SUMMARY:
This purpose of this study is to see if expanded urine culture techniques used in the laboratory improve the clinical care of women over standard urine culture techniques.

DETAILED DESCRIPTION:
The investigators request permission to recruit 225 women who respond "yes" to the question "do you feel you have a urinary tract infection". All participants will provide baseline urine specimens obtained by transurethral catheter (to avoid vulvo-vaginal contamination) and will complete a UTISA questionnaire to assess their current urinary tract symptoms. Participants will be randomized to the SUC treatment algorithm or the EQUC treatment algorithm. Treating physicians will receive either the SUC results or the EQUC results from the clinical laboratory and the results will be part of their clinical record. Treating physicians will follow the Loyola FPMRS treatment algorithm. Women in the study will also give consent for us to contact them using email, text messaging or phone call within 7-10 days after "treatment plan" has been implemented. The treatment plan options will include no treatment if the culture results show no pathogenic bacteria. All participants will be queried 7-10 days after their treatment plan (by email or text) "do you feel you continue to have a urinary tract infection". Women who respond "yes' will be asked to return for a second urine specimen which is our standard protocol. The second urine specimen will be analyzed using EQUC culture techniques only. Again, a treatment plan will be developed by the attending physician and the patient participant will be queried 7-10 days after the plan is implemented.

ELIGIBILITY:
Inclusion Criteria:

* A "yes" answer to the screening question "do you feel you have a UTI"?
* Non-pregnant women ages 18 years or older
* Agreement to respond to a text or email question 7-10 days after treatment plan for their UTI (note: the treatment plan may include "no treatment").

Exclusion Criteria:

* Women currently on antibiotics
* Patients who cannot communicate or read in English
* Patients under the age of 18
* Pregnant patients
* Women with an indwelling catheter and intermittent self-catheterization
* Men
* Urine obtained via the "clean catch method" (i.e. voided urine)
* Women who refuse to be catheterized
* Women who cannot or will not agree to respond to an email or text message 7-10 days after treatment plan is initiated.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Compare UTI symptom resolution rates in women with symptoms of UTI who are treated based on EQUC versus SUC results. | 4 weeks
  Using the FPMRS treatment algorithms (see appendix I & II Standard Urine Culture Treatment and Expanded Urine Culture Treatment Algorithms), attending physicians will treat participants based on their randomization to EQUC versus SUC. Following a 3-5 day standard course of treatment (which may include no antibiotics if the culture is negative), participants will be queried 7-10 days "do you continue to have UTI symptoms". Women who report "no" will be categorized as successful treatment, women who respond "yes" will be categorized as treatment failures.

SECONDARY OUTCOMES:
Revise the EQUC treatment algorithm. | 6 months
  The EQUC treatment algorithm was based on known uropathogens that we had previously identified as most likely to be symptomatic. During the course of this work we may identify other pathogens that are present and causing symptoms. These organisms will be identified and added to the treatment algorithm. This interim analysis is planned and was part of the statistical calculations to determine sample size.
Identify the symptom profile associated with specific organisms. | 1 year
  Using the UTISA questionnaire, we will perform a symptoms association study with specific bacteria.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Mueller, MD, Principal Investigator — Loyola University
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] KASS EH. Asymptomatic infections of the urinary tract. Trans Assoc Am Physicians. 1956;69:56-64. No abstract available. PMID 13380946
- [Result] Maskell R, Pead L, Allen J. The puzzle of "urethral syndrome": a possible answer? Lancet. 1979 May 19;1(8125):1058-9. doi: 10.1016/s0140-6736(79)92953-2. PMID 86778
- [Result] Yuan S, Cohen DB, Ravel J, Abdo Z, Forney LJ. Evaluation of methods for the extraction and purification of DNA from the human microbiome. PLoS One. 2012;7(3):e33865. doi: 10.1371/journal.pone.0033865. Epub 2012 Mar 23. PMID 22457796